CLINICAL TRIAL: NCT00096798
Title: A Double-Blind, Placebo-Controlled Study of Ethyl Eicosapentanoic Acid (Ethyl-EPA) in Major Depressive Disorder
Brief Title: Ethyl Eicosapentanoic Acid (Ethyl-EPA) for Treating Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K23AT001129 (NIH)
Record Dates: First submitted 2004-11-15; First posted 2004-11-16 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Depressive Disorder; Depression
Keywords: Fatty Acids, Omega-3; Antidepressive Agents; Eicosapentanoic Acid
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — eicosapentaenoic acid ethyl ester

INTERVENTIONS:
Drug: Ethyl-eicosapentanoic acid (ethyl-EPA)

SUMMARY:
The purpose of this study is to examine the effectiveness of ethyl-eicosapentanoic acid (ethyl-EPA), an omega-3 fatty acid, in treating depression.

DETAILED DESCRIPTION:
Evidence suggests that omega-3 fatty acids may help reduce symptoms of depression. This study will determine whether ethyl-EPA, an omega-3 fatty acid, can be used safely and effectively to treat major depression.

Participants will be randomly assigned to receive either ethyl EPA-containing pills or placebo daily for 8 weeks. Each week, participants will be asked to complete questionnaires which will be used to assess the severity of their depression.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder

Exclusion Criteria:

* Serious comorbid psychiatric disorder
* Unstable medical illness
* Prior use of any omega-3 fatty acid product

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2001-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Alleviation of depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: David Mischoulon, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851
- [Derived] Mischoulon D, Papakostas GI, Dording CM, Farabaugh AH, Sonawalla SB, Agoston AM, Smith J, Beaumont EC, Dahan LE, Alpert JE, Nierenberg AA, Fava M. A double-blind, randomized controlled trial of ethyl-eicosapentaenoate for major depressive disorder. J Clin Psychiatry. 2009 Dec;70(12):1636-44. doi: 10.4088/JCP.08m04603. Epub 2009 Aug 25. PMID 19709502